CLINICAL TRIAL: NCT03624517
Title: Comparison of 24-hours Versus 72-hours of Octreotide Infusion Along With Endoscopic Therapy in Preventing Early Rebleed From Esophageal Varices: a Multi-center, Randomized Clinical Study
Brief Title: Comparison of 24-hours Versus 72-hours of Octreotide Infusion in Preventing Early Rebleed From Esophageal Varices
Acronym: LOVARB
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment was severely affected due to COVID, so study was stopped prematurely.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Ohio State University (Other); University of Texas Southwestern Medical Center (Other); University of Florida Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00027015
Record Dates: First submitted 2018-07-31; First posted 2018-08-10 (Actual); Results first posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Varices; Liver Cirrhoses; Bleeding Esophageal Varices; Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Esophageal and Gastric Varices; Gastrointestinal Hemorrhage | interventions — Octreotide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 24-hour octreotide infusion (Experimental): Patients will receive octreotide infusion over 24 hours
  Interventions: Drug: Octreotide
- 72-hour octreotide infusion (Active Comparator): Patients will receive octreotide infusion over 72 hours
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Octreotide — Octreotide infusion for 24-hours in patients with bleeding esophageal varices.

SUMMARY:
This study evaluates the safety and efficacy of 24-hour vs 72-hour octreotide infusion after variceal banding in cirrhotic patients with bleeding esophageal varices.

DETAILED DESCRIPTION:
In cirrhotic patients with bleeding esophageal varices, standard of care therapy includes administration of octreotide infusion over 72-hours and endoscopic banding of esophageal varices.

Octreotide acts to reduce the pressure in the blood vessels surrounding the liver, decreasing the propensity of bleeding from esophageal varices. The recommended duration of octreotide therapy is based largely on expert opinion, however a 72-hour duration of treatment is likely to be unnecessary and may inappropriately increase hospital and medical costs.

This study aims to determine the safety of 24-hours of octreotide infusion in patients with bleeding esophageal varices.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females who are 18 years of age or older.
2. Evidence or suspicion of upper gastrointestinal bleed (GIB)
3. Patient with known or suspected cirrhosis
4. Upper GIB secondary to bleeding esophageal varices as show by esophageal endoscopy, requiring endoscopic band ligation (EBL) at presentation
5. Willing and able to provide informed consent for study, or have a Legally authorized representative (LAR) provide consent if the patient is unable to do so

Exclusion Criteria:

1. Known upper gastrointestinal malignancy
2. Bleeding from gastric varices, with or without esophageal varices
3. Use of any other endoscopic method to stop GI bleeding beyond endoscopic band ligation
4. Variceal bleeding in the last 90 days
5. History of transjugular, intrahepatic, portosystemic shunt (TIPS) or vascular decompression surgery
6. Pregnant females
7. Incarcerated individuals
8. Myocardial infarct, cerebrovascular accident, sepsis, respiratory failure, or severe intercurrent illness within the previous 6 weeks
9. Non-cirrhotic portal hypertension causing esophageal varices
10. Known or suspected allergy to octreotide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Rockey, M.D, Principal Investigator — Medical University of South Carolina
Locations (8):
- United States (8):
  - University of Florida Health, Jacksonville, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - The Ohio state University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas at Austin, Austin, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Brooke Army Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Allam J, De Melo S, Feagins LA, Agrawal D, Malespin M, Shuja A, Lara LF, Rockey DC. Comparison of 24 vs 72-hr octreotide infusion in acute esophageal variceal hemorrhage - A multi-center, randomized clinical trial. Am J Med Sci. 2025 Jan;369(1):71-76. doi: 10.1016/j.amjms.2024.08.027. Epub 2024 Sep 4. PMID 39241828

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 24-hour octreotide infusion | 72-hour octreotide infusion
Started | 15 | 19
Completed | 15 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 24-hour Octreotide Infusion | 72-hour Octreotide Infusion | Total
Number analyzed (Participants) | 15 | 19 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (16) | 54 (11) | 53.12 (13.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 8 | 13 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 11 | 16 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 15 | 19 | 34

OUTCOME MEASURES:

1. Primary Outcome: Esophageal Varices Rebleed Within 72-hours After Control of Initial Bleed
Description: Rebleeding within 72-hours will be defined as any of the following:
  1. A drop in hemoglobin by more than 20 percentage points from baseline
  2. Sustained tachycardia above 100 beats per minute, with or without hematochezia or melena
  3. Transfusion of >2 unites packed red blood cells after esophageal band ligation
  4. Recurrence of hematemesis or ongoing melena
  5. Urgent or emergent need for Transjugular Intrahepatic Portosystemic Shunt (TIPS) to control suspected rebleeding
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 24-hour octreotide infusion | 72-hour octreotide infusion
Number analyzed (Participants) | 15 | 19
Participants | 0 | 1

2. Secondary Outcome: Esophageal Varices Rebleed at 7 Days and 30 Days After Control of Initial Bleed
Description: Rebleeding after 72-hours will be defined as:
  1. Any new episode of hematemesis, melena, or hematochezia (with hemodynamic instability)
  2. Drop in hemoglobin by more than 20 percentage points OR the need for >2 units packed red blood cells
  3. Need for TIPS or surgery to control suspected bleeding
Time Frame: 7 days and 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 24-hour octreotide infusion | 72-hour octreotide infusion
Number analyzed (Participants) | 15 | 19
Participants
  Rebleeding at 7 Days | 0 | 1
  Rebleeding at 30 Days | 0 | 2

3. Secondary Outcome: Survival at 7 Days and 30 Days After Control of Initial Bleed
Description: Survival at 7 days and 30 days.
Time Frame: 7 days and 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 24-hour octreotide infusion | 72-hour octreotide infusion
Number analyzed (Participants) | 15 | 19
Participants
  Survival at 7 Days | 15 | 19
  Survival at 30 Days | 15 | 18

ADVERSE EVENTS:
Time Frame: up to 30 days
Arm/Group | 24-hour octreotide infusion | 72-hour octreotide infusion
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/19
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/19
Other Adverse Events (participants affected / at risk) | 2/15 | 8/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24-hour octreotide infusion (N=15) | 72-hour octreotide infusion (N=19)
Death (Sepsis) (General disorders) | 0 (0) | 1 (1) — Sepsis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24-hour octreotide infusion (N=15) | 72-hour octreotide infusion (N=19)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Dysphagia/Odynophagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nasogastric Tube Insertion (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mechanical Ventilation >12h (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Vasopressor Use (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT03624517/Prot_SAP_000.pdf